CLINICAL TRIAL: NCT05135858
Title: Dose Dense Re-challenge of High Dose Methotrexate (HD-MTX) With Glucarpidase (CPG2) for Relapsed Primary Central Nervous System Lymphoma (PCNSL): A Phase I Trial
Brief Title: Dose Dense Re-challenge of High Dose Methotrexate With Glucarpidase for Relapsed Primary Central Nervous System Lymphoma
Acronym: METHOGLU
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APHP201186; 2021-000210-42 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2021-11-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary CNS lymphoma; Relapse; High-dose methotrexate; Glucarpidase
MeSH Terms: conditions — Recurrence | interventions — glucarpidase; Methotrexate

STUDY DESIGN:
Intervention Model Description: The phase I will follow a standard "3+3" dose level escalation design with reduced time interval of HD-MTX injections at fixed dose of HD-MTX to establish the minimum tolerated time interval.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPG2 (Experimental): 6 infusions of glucarpidase
  Interventions: Drug: Glucarpidase; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Glucarpidase — Glucarpidase (CPG2) Dose: 2000 U (2 vials of 1000 U per dose) 5 minutes-intravenous administration 24 hours after each Methotrexate infusion (i.e. 6 times in the whole protocol)
Drug: Methotrexate (MTX) — MTX will be administred 6 times during the protocol, at a variable interval of 8, 6 or 5 days. It will be administrated in a 2 to 3-hour IV infusion, at the dose of 3.5 g/m2 (body surface area capped at 2 m2). Each MTX administration will be preceded by a prehydration and will be followed by a posthydration

SUMMARY:
High dose intravenous Methotrexate (HD-MTX) is the key drug in the treatment of primary central nervous system lymphoma (PCNSL). HD-MTX is usually delivered with time interval ranging from 10 to 21 days. Reduction of injection time interval is limited by MTX renal excretion and systemic toxicity.

Glucarpidase (CPG2) is a recombinant bacterial rescue enzyme that cleaves circulating MTX into inactive metabolites, reducing plasma MTX concentrations within few minutes.

The research hypothesis is that CPG2 used after HD-MTX injection allows to reduce time interval between MTX injections, increase dose intensity of the chemotherapy, reduce systemic toxicity and duration of hospitalization.

DETAILED DESCRIPTION:
Open-label multicenter Phase I dose finding trial based on 3+3 escalation design. The phase I will follow a standard "3+3" dose level escalation design with reduced time interval of HD-MTX injections at fixed dose of HD-MTX to establish the minimum tolerated time interval.

HD-MTX (methotrexate) is administered intravenously at the dose 3.5 g/m² (body surface area capped at 2 m2) over 2 to 3 hours, followed at H24 by glucarpidase with a 3 different MTX administration intervals: 8 days, 6 days, and 5 days.

Treatments will be continued for a maximum of 6 injections until disease progression, unacceptable toxicity, or investigator's/patient's decision.

Three dose levels could be explored under toxicity restrictions, where the dose combination for each cohort of three subjects will be determined by 3+3 escalation rule. Three schedule dose levels will be : every 8 days, every 6 days and every 5 days.

The starting schedule dose of HD-MTX will be one administration of HD-MTX every 8 days for 6 injections.

Dose of MTX will be fixed and will not be modified. No skipping of the dose level will be allowed. No intra-patient dose escalation is allowed.

The DLT evaluation period begins with the first dose of methotrexate and ends at the beginning of the 25th day after the first MTX infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral relapse of primary CNS lymphoma (any line)
2. Pathological diagnosis of diffuse large B cell lymphoma (or cytological diagnosis in the CSF or in the vitreous) at initial diagnosis (not mandatory at the time of the present relapse)
3. Absence of any systemic involvement confirmed by full body CT scan and/or FDG-PET scan
4. Age≥18 years
5. HD-MTX based chemotherapy in first line treatment, with complete response lasting at least 6 months after the end of the 1st line treatment
6. No administration of other anticancer therapy within the 3 weeks prior to inclusion
7. Karnofsky performance status (KPS) ≥ 50
8. Adequate haematological, renal and hepatic function (adequate Laboratory Parameters within 21 days):

   1. Absolute neutrophil count (ANC) >1000/mm3
   2. Platelets > 100,000/mm3 independent of transfusion support
   3. Alanine aminotransferase and aspartate aminotransferase ≤ 3 x upper limit of normal (ULN) and/or total bilirubin ≤ 1,5x ULN, unless related to Gilbert's or Meulengracht disease
   4. Estimated Glomerular Filtration Rate ≥ 60 mL/min/1.73m2) (MDRD)
9. All non-hematological adverse events (AEs) related to prior therapy completely resolved or improved to Grade 1-2 (except for alopecia or fatigue).
10. Written informed consent, which could be signed by the trustworthy person or close relatives in case the neurologic status of the patient does not allow him to sign. In case the patient is unable to sign the consent at baseline, but his neurological status improves during the treatment, he will be asked to give his written informed "follow-up" consent

Exclusion Criteria:

1. Positive HIV serology
2. Active viral infection with Hepatitis B or C virus
3. Preexisting immunodeficiency (organ transplant recipient)
4. Relevant congestive heart failure interfering with hydration
5. Isolated CNS relapse of systemic non-Hodgkin's lymphoma (NHL)
6. Pregnancy or lactation. An effective contraception is mandatory for patients (men and women of childbearing potential) all along the study participation and during at least 6 months after the end of MTX. Men must not donate sperm all along the study participation and during at least 6 months after the end of MTX.
7. Third space (i.e. pleural effusion, ascites, extended oedema).
8. Obesity (body mass index >30 kg/m2).
9. Any other active malignancy, except basocellular carcinoma and non-invasive cervix cancer
10. Absolute contraindication to MTX or leucovorin
11. Previous use of carboxypeptidase for delayed MTX excretion and kidney dysfunction after HD-MTX
12. No social security affiliation
13. Persons under legal protection (tutorship or curatorship) or safety measure
14. Participation in any other clinical trial (Jardé 1 and 2) either 1 month prior to or during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of a dose schedule limiting toxicity (DLT) | 25th day after the first injection of methotrexate
  defined as any of the following events assessed as related or possibly related to methotrexate:
  * Any grade V toxicity (according to NCI-CTCAE v 5.0)
  * Grade IV non-haematological toxicity excluding fatigue, alopecia, nausea, vomiting (according to NCI-CTCAE v 5.0)
  * Creatinine > 3 X baseline (grade III toxicity according to NCI-CTCAE v 5.0)
  * Grade IV thrombopenia, grade III thrombopenia with bleeding, grade IV neutropenia or grade III neutropenia with fever,lasting > 3 days (according to NCI-CTCAE v 5.0)
  * Delay in MTX administration > 36 hours due to any adverse effect.

SECONDARY OUTCOMES:
Frequency and grading of adverse event according to NCI-CTCAE v5.0 | through study completion, an average of 4 months
Mean score of neurocognition assessed by neuropsychological testing at baseline and within the - Neurocognition assessed by neuropsychological testing at baseline and within the 3 months after the end of HD-MTX treatment | 3 months after the end of HD-MTX treatment
Overall response rate according to IPCG criteria | After 3 cycles (each cycle is 5, 6 or 8 days), at the end of treatment (up to 48 days) and at 3 months after the end of treatment (up to 48 days)
Mean of dosages of MTX and its metabolites in the blood, urine and cerebrospinal fluid (CSF) | At the first and the third cycles (each cycle is 5, 6 or 8 days)
Mean of dosage of anti-glucarpidase antibodies | At baseline, then prior to each CPG2 dose, at the end of HD-MTX treatment (up to 48 days) and at 3 months after the end of HD-MTX treatment.(up to 48 days)
Mean global score of quality of life assessment measured with EORTC QLQ-C30 scale | At baseline, at the end of HD-MTX treatment (up to 48 days) and at 3 months after the end of HD-MTX treatment (up to 48 days)]
Mean global score of quality of life assessment measured with Brain Module (BM 20) | At baseline, at the end of HD-MTX treatment (up to 48 days) and at 3 months after the end of HD-MTX treatment (up to 48 days)
Median duration of treatment-related hospitalization in acute care unit | From day 1 until discharge from hospital, an average of 4 to 7 weeks
  Defined as the cumulative time from start of the HD MTX protocol (including the pre-hydration) to its elimination
Mean of dosage of CSF IL-10 | At baseline and at the end of the treatment (up to 48 days)
Median duration of hospitalization during the treatment | From day 1 until end of the treatment (up to 48 days)
  Duration of treatment-related hospitalization in acute care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.